CLINICAL TRIAL: NCT05371067
Title: Fructose Effect on Neuroinflammation and Feelings: Direct Action on the Brain or Indirect by the Intestinal Microbiota?
Brief Title: Fructose Effect on Neuroinflammation and Feelings
Acronym: MOODYFRUCTOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/0209/HP
Record Dates: First submitted 2022-01-03; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-01

CONDITIONS: Gastro-Intestinal Disorder
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: This study is a monocentric, prospective, non-randomized, comparative assay in which volontarees are enrolled in order to study the fructose effects on intestinal microbiote and their consequencies on the emotions and the neuroinflammation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Other)
  Interventions: Other: Fructose respiratory test

INTERVENTIONS:
Other: Fructose respiratory test — Healthy volunteers will performed a fructose respiratory test in order to evaluate if they are or not fructose malabsorbing. The two population will be compared about their feelings and their micriobiote.

SUMMARY:
Fructose is increasingly present in our food. The increase in its consumption is associated with the increase in the prevalence of several pathologies such as metabolic syndrome or hepatic steatosis. The effect of fructose consumption on brain health has been poorly studied. Studies in animal models show that diets enriched in fructose promote the development of emotional behavior disorders. Fructose malabsorption is also associated with changes in the microbiota that could also impact brain health. However, no human study to date has associated fructose malabsorption with changes in the gut microbiota and effects on brain health.

The objective of this study is to study the emotional behavior of a population of healthy volunteers according to the presence or not of fructose malabsorption. Patients with fructose malabsorption are susceptible to gut dysbiosis without necessarily consuming high amounts of fructose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18 to 35
* Male sex
* BMI between 18.5 and 25
* Affiliation to a social security scheme
* Adult patient having read and understood the information letter and signed the consent form

Exclusion Criteria:

* Presence of irritable bowel syndrome, celiac disease
* Presence of a psychiatric illness
* Presence of a neurodegenerative disease
* Presence of an eating disorder
* Presence of chronic disease, including inflammatory disease
* Presence of diabetes
* Presence of an acute infectious disease
* Presence of a surgical history of the digestive tract (excluding appendectomy)
* Taking long-term treatment
* Taking antibiotics within 6 months
* Taking probiotics within 3 months
* Typical diet low in lactose, FODMAP, gluten, vegetarian, vegan, vegan, chromonutrition .... in progress
* Smoker
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection / under guardianship or guardianship
* Simultaneous participation in another interventional clinical trial

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-08-08 (Estimated); Study Completion 2022-08-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the chronic effect of fructose on anxiety in healthy volunteers with fructose malabsorption compared to healthy volunteers without fructose malabsorption. | At the inclusion visit (V1)
  Spielberger State Anxiety Questionnaire Score (STAI)

SECONDARY OUTCOMES:
Evaluate the fructose consumption in healthy volunteers with fructose malabsorption compared to healthy volunteers without fructose malabsorption. | For 7 days before V2
  Usual fructose consumption assessed by dietary log over 7 days
Evaluate the chronic effect of fructose on depression in healthy volunteers with fructose malabsorption compared to healthy volunteers without fructose malabsorption. | At the inclusion visit (V1)
  HAD score
Evaluate the chronic effect of fructose on low-grade intestinal inflammation in healthy volunteers with fructose malabsorption compared to healthy volunteers without fructose malabsorption. | up to 1 month
  Score STAI
Evaluate the chronic effect of fructose on microbiota's composition in healthy volunteers with fructose malabsorption compared to healthy volunteers without fructose malabsorption. | up to 1 month
  Amplicon sequencing of the V3-V4 area (region) of bacterial 16S rRNA in volunteer's faeces

CONTACTS AND LOCATIONS:
Overall Officials: Chloé Melchior, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU de ROUEN, Rouen, France